CLINICAL TRIAL: NCT01274559
Title: A Worldwide, Multicenter, Double-Blind, Randomized, Parallel, Placebo-Controlled 12-Week Study to Evaluate the Efficacy and Safety of Extended Release (ER) Niacin/Laropiprant When Added to Ongoing Lipid-Modifying Therapy in Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia
Brief Title: Efficacy and Safety of Extended Release (ER) Niacin/Laropiprant When Added to Ongoing Lipid-Modifying Therapy in Patients With High Cholesterol or Abnormal Lipid Levels (MK-0524A-133)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: In HPS2-THRIVE, MK-0524A did not meet the primary efficacy objective and there was a significant increase in incidence of some types of non-fatal SAEs
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-133; CTRI/2012/08/002857 (Registry Identifier: CTRI); 2010-021627-27 (EudraCT Number)
Record Dates: First submitted 2010-10-25; First posted 2011-01-11 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemia
Keywords: MK-0524A/ER; Hypercholesterolemia; Dyslipidemia; Niacin; Laropiprant
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended-release niacin/laropiprant (Experimental): ERN/LRPT 1 g (1 tablet for 4 wks) followed by ERN/LRPT 2 g (2 tablets for 8 wks); Each 1-g tablet contains 1 g of ER niacin and 20 mg of laropiprant.
  Interventions: Drug: Extended-release niacin/laropiprant (ERN/LRPT)
- Placebo (Placebo Comparator): Matching 1 g Placebo (1 tablet for 4 wks) followed by 2 g placebo (2 tablets for 8 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Extended-release niacin/laropiprant (ERN/LRPT) — 1 oral 1 g tablet of ERN/LRPT to be taken with food in the evening or at bedtime for the first 4 weeks of treatment; then 2 oral 1g tablets of ERN/LRPT to be taken together in the evening or at bedtime with food for the next 8 weeks. Each 1g tablet contains 1g ERN and 20 mg LRPT
  Arms: Extended-release niacin/laropiprant
Drug: Placebo — 1 oral 1 g tablet of placebo to be taken with food in the evening or at bedtime for the first 4 weeks of treatment; then 2 oral 1g tablets of placebo to be taken together in the evening or at bedtime with food for the next 8 weeks.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study in participants with primary hypercholesterolemia or mixed dyslipidemia, and elevated low density lipoprotein-cholesterol (LDL-C) to assess the efficacy and safety of extended release (ER) niacin/laropiprant [ERN/LRPT (MK-0524A)] when added to the following ongoing lipid-modifying therapy (LMT): simvastatin,

atorvastatin, rosuvastatin monotherapy, ezetimibe/simvastatin fixed dose combination (FDC), or any statin co-administered with ezetimibe. The study is based on the hypothesis that ERN/LRPT 2 g daily will be superior to placebo at lowering LDL-C at Week 12 of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has a history of primary hypercholesterolemia or mixed dyslipidemia.
* Must meet one of the risk categories (very high, high or moderate and corresponding LDL-C criteria at Visit 2.
* Has TG levels <500 mg/dL (<5.65 mmol/L).
* Has been on a stable dose of one of the following lipid-modifying therapies (LMTs)for at least 6 weeks prior to Visit 1, and agrees to remain on the same type and dose of LMT for the duration of the study:

  * Monotherapy: any statin
  * Combination Therapy: ezetimibe/simvastatin in the same tablet
  * Co-administration Therapy: any statin co-administered with ezetimibe
* Is male or female and ≥18 years of age on day of signing informed consent.
* A female must meet ONE of the following:

  * Of reproductive potential and agrees to remain abstinent or use (or have their partner use) 2 acceptable methods of birth control for the study duration.
  * Not of reproductive potential is eligible without requiring the use of contraception. Definition of "not of reproductive potential": one who has either of the following:

    * reached natural menopause, defined as: 6 months of spontaneous amenorrhea with serum FSH levels (at Visit 1) in the postmenopausal range (per central lab) or 12 months of spontaneous amenorrhea.Spontaneous amenorrhea does not include cases for which there is an underlying disease that causes amenorrhea (e.g., anorexia nervosa).
    * 6 weeks post surgical hysterectomy, or bilateral oophorectomy with or without hysterectomy.
    * Bilateral tubal ligation without subsequent restorative procedure.
* Understands the study's procedures, alternative treatments available, risks involved with the study, and voluntarily agrees to participate by giving written informed consent.

Exclusion Criteria

- Has taken a prohibited LMT within 6 weeks of Visit 1. Examples of

prohibited LMT include bile acid sequestrants, fibrates (monotherapy, coadministration or combination with other LMT), niacin >50 mg, and red yeast rice products.

* Has had a change to the type or dose of acceptable LMT regimen within 6 weeks of Visit 1.
* Is pregnant, breastfeeding, or expecting to conceive during the study including the 14-day poststudy follow-up.
* Has a history of malignancy ≤5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Female who is expecting to donate eggs during the study, including the 14-day follow-up.
* Is unlikely to adhere to the study procedures, keep appointments, or is planning to relocate during the study.
* Has participated in a study, including post-study follow-up, with an investigational compound (non-lipid-modifying) within 30 days of Visit 1 or a lipid-modifying compound (investigational or marketed), within 6 weeks of Visit 1.
* Has donated and/or received blood as follows:

  * donated blood products or has had phlebotomy of >300 mL within 8 weeks prior to signing informed consent.
  * intends to give or receive blood products during the study.
  * intends to donate more than 250 mL of blood products within 8 weeks following the last study visit.
* Has the following exclusionary laboratory values at Visit 2

  * Creatinine clearance (eGFR) <30 mL/min (0.50 mL/s)
  * ALT (SGPT) >1.5 x ULN
  * AST (SGOT) >1.5 x ULN
  * CK >2 x ULN
* Has used recreational or illicit drugs within 1 year of signing informed consent.
* Was <80% compliant with LMT or placebo at Visit 2, AND in the opinion of the investigator, is believed to be unable to maintain at least 80% compliance with dosing during the active treatment period.
* Has chronic heart failure defined by the New York Heart Association (NYHA) Classes III or IV, uncontrolled cardiac arrhythmias, or poorly controlled hypertension (systolic blood pressure >160 mm Hg or diastolic >100 mm Hg).
* Has Type 1 or Type 2 diabetes mellitus and meets one or more of the following criteria:

  * Is poorly controlled (HbA1C >8.0% at Visit 1)
  * Is newly diagnosed (within 3 months of Visit 1)
  * Has recently experienced repeated hypoglycemia or unstable glycemic control (within 3 months of Visit 1).
  * Is taking new or recently adjusted antidiabetic pharmacotherapy (with the exception of ± ≤ 10 units of insulin) within 3 months of Visit 1.
* Has uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins (i.e., secondary causes of hyperlipidemia such as hyper- or hypothyroidism.
* Has nephrotic syndrome or other clinically significant renal disease.
* Has active peptic ulcer disease within 3 months of Visit 1.
* Has a history of hypersensitivity or allergic reaction to niacin or niacin containing products.
* Has history of myocardial infarction, stroke, coronary artery bypass surgery or other revascularization procedure, unstable angina or angioplasty within 3 months of Visit 1.
* Has arterial bleeding.
* Has a history of ileal bypass, gastric bypass or other significant condition associated with malabsorption or rapid weight loss within 18 months of Visit 1.
* Has active or chronic hepatobiliary or hepatic disease.
* Is Chinese and is on simvastatin 80 mg or a product containing simvastatin 80 mg at Visit 1.
* Is receiving treatment with systemic steroids (intravenous, injected, and oral steroids) OR systemic anabolic agents.
* Consumes more than 3 alcoholic drinks on any given day or more than 14 drinks per week.
* Is taking the following antioxidant vitamins each day:

  * Vitamin C in excess of 1500 mg
  * Vitamin E in excess of 45 IU for men, 36 IU for women
  * Beta Carotene 15000 IU for men, 12000 IU for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1173 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2013-02-26 (Actual); Study Completion 2013-02-26 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0524A-133&kw=0524A-133&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 3 study HPS2-THRIVE (NCT00461630) did not meet its primary endpoint of reduction of major vascular events and had a significant increase in the incidence of some types of non-fatal serious adverse events. As a result, MK-0524A-133 was discontinued. Only individual data were obtained; none of the planned efficacy outcomes were summarized.
Groups:
- Extended-release Niacin/Laropiprant: Extended-release niacin (ERN)/laropiprant (LRPT) 1 g (1 tablet for 4 wks) followed by ERN/LRPT 2 g (2 tablets for 8 wks); Each 1-g tablet contains 1 g of ER niacin and 20 mg of laropiprant.
Period: Overall Study
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Started | 587 | 586
Treated | 572 | 572
Completed | 390 | 441
Not Completed | 197 | 145
Not completed — Adverse Event | 57 | 13
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 3 | 3
Not completed — Non-compliance with Study Drug | 2 | 4
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 28 | 23
Not completed — Study Terminated by Sponsor | 79 | 87
Not completed — Withdrawal by Subject | 25 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended-release Niacin/Laropiprant | Placebo | Total
Number analyzed (Participants) | 587 | 586 | 1173
Age, Customized [Number; unit: Participants]
  21 to 30 years | 1 | 2 | 3
  31 to 40 years | 9 | 12 | 21
  41 to 50 years | 63 | 62 | 125
  51 to 60 years | 182 | 168 | 350
  61 to 70 years | 209 | 232 | 441
  71 to 80 years | 108 | 98 | 206
  >80 years | 15 | 12 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239 | 243 | 482
  Male | 348 | 343 | 691

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline at Week 12 in Low Density Lipoprotein-Cholesterol (LDL-C)
Time Frame: Baseline and Week 12
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percent Change From Baseline in LDL-C:High-density Lipoprotein Cholesterol (HDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percent Change From Baseline in Triglyceride (TG) at Week 12
Time Frame: Baseline and Week 12
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B) at Week 12
Time Frame: Baseline and Week 12
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percent Change From Baseline in Apo B:Apolipoprotein A-I (Apo A-I) at Week 12
Time Frame: Baseline and Week 12
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC):HDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percent Change From Baseline in Lipoprotein a [Lp(a)] at Week 12
Time Frame: Baseline and Week 12
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percent Change From Baseline in Apo A-I at Week 12
Time Frame: Baseline and Week 12
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percent Change From Baseline in TC at Week 12
Time Frame: Baseline and Week 12
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percent Change From Baseline in LDL-C at Week 4
Time Frame: Baseline and Week 4
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Percent Change From Baseline in LDL-C:HDL-C at Week 4
Time Frame: Baseline and Week 4
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 4
Time Frame: Baseline and Week 4
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Percent Change From Baseline in TG at Week 4
Time Frame: Baseline and Week 4
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 4
Time Frame: Baseline and Week 4
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Percent Change From Baseline in Apo B at Week 4
Time Frame: Baseline and Week 4
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Percent Change From Baseline in Apo B:Apo A-I at Week 4
Time Frame: Baseline and Week 4
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Percent Change From Baseline in TC:HDL-C at Week 4
Time Frame: Baseline and Week 4
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Percent Change From Baseline in Lp(a) at Week 4
Time Frame: Baseline and Week 4
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Percent Change From Baseline in Apo A-I at Week 4
Time Frame: Baseline and Week 4
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Percent Change From Baseline in TC at Week 4
Time Frame: Baseline and Week 4
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Number of Participants Who Achieve LDL-C Target Levels at Week 12 of Treatment
Description: assessed as per National Cholesterol Education Program (NCEP) Adult Treatment Panel III (ATP III) and European Society of Cardiology (ESC) treatment guidelines
Time Frame: Baseline and 12 weeks
Population: Study was terminated. Efficacy endpoints were not summarized and no planned efficacy analyses were performed.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Description: The All Patients as Treated (APaT) population, which consisted of all randomized participants who received at least one dose of study treatment post randomization.
Arm/Group | Extended-release Niacin/Laropiprant | Placebo
Serious Adverse Events (participants affected / at risk) | 23/572 | 16/572
Other Adverse Events (participants affected / at risk) | 101/572 | 16/572
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended-release Niacin/Laropiprant (N=572) | Placebo (N=572)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Puncture site infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 1 (1)
Diabetic macroangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended-release Niacin/Laropiprant (N=572) | Placebo (N=572)
Pruritus (Skin and subcutaneous tissue disorders) | 45 (52) | 3 (3)
Flushing (Vascular disorders) | 66 (100) | 13 (18)

LIMITATIONS AND CAVEATS:
MK-0524A-133 was stopped prior to completion. Raw individual efficacy data were obtained but none of planned efficacy outcomes were summarized or analyzed. Only safety data were summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.